CLINICAL TRIAL: NCT06321211
Title: Development of a Novel Asian Mediterranean Diet and Its Acceptability in Non- Alcoholic Fatty Liver Disease (NAFLD)- a Pre-intervention Study
Brief Title: Development of a Novel Asian Mediterranean Diet and Its Acceptability in NAFLD
Acronym: aMed
Status: Active, not recruiting | Type: Observational
Sponsor: Singapore Institute of Technology (Other)
Collaborators: Singapore Health Services (Other)
Responsible Party: Principal Investigator, Verena Tan Ming Hui, Associate Professor, Singapore Institute of Technology
Other Study IDs: RECAS-0244
Record Dates: First submitted 2024-02-29; First posted 2024-03-20 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Fatty Liver, Nonalcoholic
Keywords: Mediterranean Diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this pre-intervention study is test the acceptability of Asian version of the Mediterranean diet to NAFLD patients.

The main question[s] it aims to answer are:

1. Whether Asian version of the Mediterranean diet that retains the nutritional composition and can be developed by mapping the components of the Mediterranean diet and finding substitute ingredients commonly eaten in Southeast Asia.
2. Whether the 4-week menu cycle of newly developed novel Asian Mediterranean diet is acceptable among Singaporean local population.

Participants will participate in taste test sessions to find out if the Asian Mediterranean diet meals are acceptable to people with NAFLD.

DETAILED DESCRIPTION:
Numerous studies have shown that Mediterranean diet decrease the risk of cardiovascular disease, metabolic syndrome, cancer and overall mortality characterized by being low in saturated fats and animal protein, high in antioxidants, fibre and monounsaturated fatty acids, and with an adequate omega-3 to omega-6 fatty acid balance.

Recent studies have proved that adherence to a Mediterranean diet is beneficial for non-alcoholic fatty liver disease (NAFLD) as it provides antioxidants and anti-inflammatory nutrients that slows the development of hepatic steatosis.

However, adhering to the Mediterranean diet can be difficult for people of Southeast Asian cultural backgrounds to follow, as food items used in traditional Mediterranean diets may not be readily available or frequently used in local cuisines.

It is therefore the aim of this study to first map out the nutritional composition of the traditional Mediterranean diet, derive substitute ingredients, and then develop an Asian version of the Mediterranean diet that can be accepted and easily adopted by the Asian population while retaining the beneficial nutritional characteristics.

Following this, NAFLD patients will be recruited for the sensory evaluation of the Asian Mediterranean diet. Specifically for this study, the researchers are keen to focus on a clinical condition (i.e. NAFLD) that has been demonstrated to reap positive effects from adopting a Mediterranean diet. As such, this is a pre-intervention study with a focus on development and evaluating its acceptability among NAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD, as determined clinically by imaging evidence of hepatic steatosis on ultrasound/CT/MRI

Exclusion Criteria:

* Secondary causes of NAFLD (e.g. medication-induced)
* Unstable body weight (variation >5% within the preceding 3 months)
* Current use of weight loss medications
* Other liver diseases (viral hepatitis, auto-immune or cholestatic liver disease, Wilson's disease, hemochromatosis, alpha-1 anti-trypsin deficiency)
* Unstable diabetes (HbA1c >8.5%)
* Renal failure
* Inability to provide informed consent
* Pregnancy and lactation
* Problems with tasting and smelling
* Food allergy/intolerances/restrictions

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We plan to recruit adults diagnosed with NAFLD (outpatients) from the Department of Hepatology in Singapore General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
Sensory Evaluation Test Score NAFLD | 15 April to 27 Dec 2024
  Score of sensory evaluation test to assess the acceptability of Asian Mediterranean diet in subjects with NAFLD on a 7-point Likert scale. Lower score on the 7-point Likert scale of 1 to 7 (1 = Like Very Much, 7 = Dislike Very Much) would mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Verena Tan, Ph.D, Principal Investigator — +65 9172 4062
Locations (1):
- Singapore Institute of Technology, Singapore, Singapore

REFERENCES:
- [Background] Anania C, Perla FM, Olivero F, Pacifico L, Chiesa C. Mediterranean diet and nonalcoholic fatty liver disease. World J Gastroenterol. 2018 May 21;24(19):2083-2094. doi: 10.3748/wjg.v24.i19.2083. PMID 29785077
- [Background] Romero-Gomez M, Zelber-Sagi S, Trenell M. Treatment of NAFLD with diet, physical activity and exercise. J Hepatol. 2017 Oct;67(4):829-846. doi: 10.1016/j.jhep.2017.05.016. Epub 2017 May 23. PMID 28545937
- [Background] Abenavoli L, Greco M, Milic N, Accattato F, Foti D, Gulletta E, Luzza F. Effect of Mediterranean Diet and Antioxidant Formulation in Non-Alcoholic Fatty Liver Disease: A Randomized Study. Nutrients. 2017 Aug 12;9(8):870. doi: 10.3390/nu9080870. PMID 28805669

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT06321211/Prot_SAP_000.pdf
  • Informed Consent Form: Consent Form Only (2024-03-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT06321211/ICF_001.pdf
  • Informed Consent Form: Participant Information Sheet (2024-03-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT06321211/ICF_002.pdf